CLINICAL TRIAL: NCT01402388
Title: Effect of Intensive Lifestyle Intervention on Hormonal Factors Regulating Food Intake and Blood Glucose Control in Patients With New Onset Type 2 Diabetes.
Brief Title: Lifestyle Intervention in Patients With New Onset Type 2 Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Bournemouth Hospital (Other)
Responsible Party: Professor David Kerr, Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07/H0201/100
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle intervention group. (Experimental)
  Interventions: Behavioral: Group lifestyle programme

INTERVENTIONS:
Behavioral: Group lifestyle programme

SUMMARY:
The study seeks to establish if weight loss achieved through a program of intensive lifestyle management can result in improvements in GLP-1 and glycaemic control, in patients with newly diagnosed type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* New onset type 2 Diabetes
* Body mass index 25 and above
* Able to give informed consent

Exclusion Criteria:

* Hypoglycaemic and antiobesity agents, or any other prescription medication that may interfere with study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Lifestyle impact on GLP-1, HbA1c and fasting glycaemia. | 8 months following commencement of study.